CLINICAL TRIAL: NCT07189533
Title: SENior PRIorat: Ciencia Participativa Para la Mejora de Los Estilos de Vida, la Calidad de Vida, el Bienestar Emocional y Las Capacidades Locomotoras de Las Personas Mayores Del Priorat
Brief Title: SENior PRIorat: Participatory Research for the Improvement of Lifestyles, Quality of Life, Emotional Well-being, and Locomotor Abilities of Older Adults in the Priorat
Acronym: SENPRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Consell Comarcal del Priorat (Unknown); Fundación Española para la ciencia y la tecnologia (Unknown)
Responsible Party: Principal Investigator, Elisabet Llauradó, Doctor, Lecturer, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 010/2025; FCT-24-19957 (Other Grant/Funding Number: FUNDACION ESPAÑOLA PARA LA CIENCIA Y LA TECNOLOGIA (FECYT))
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Lifestyle
Keywords: Participatory research; healthy lifestyle; quality of life; older adults; rural environment

STUDY DESIGN:
Intervention Model Description: Intervention group: receive the co-created intervention Control group: still with habitual lifestyle.
Who Masked: Outcomes Assessor
Masking Description: The allocation will not be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive the co-created intervention
  Interventions: Behavioral: Co-created intervention
- Control (No Intervention): still with their habitual lifestyle

INTERVENTIONS:
Behavioral: Co-created intervention — Intervention generated by a participatory research process (co-creation) in the elderly population living in rural areas to co-create solutions to improve their lifestyles, quality of life and health.
  Arms: Intervention

SUMMARY:
Spain is experiencing a demographic shift towards an ageing population. In 2022, 20.1% of Spaniards were 65 or older, a figure projected to reach 30.4% by 2050. The trend is especially marked in rural areas, where outmigration of younger generations has left a high concentration of older residents. In Catalonia's Priorat county, the share of people aged 65+ already exceeds 20%, reaching 30%, and even 40% in some villages.

The ageing process brings biological changes that reduce locomotor and cognitive abilities, limiting autonomy and quality of life. In rural areas, these challenges are compounded by social isolation and the lack of support networks, making older adults more vulnerable. Healthy lifestyle habits-such as balanced nutrition, regular exercise, avoiding tobacco and alcohol, and good sleep-can help delay dependence, lower the risk of chronic disease, and improve well-being. To promote these habits, social innovation must generate new services and approaches that address real needs, barriers, and motivations in adopting healthier lifestyles.

Our group's research shows that participatory science is an effective tool to promote healthy ageing in rural settings. A three-month intervention co-designed with older adults in villages of ≤2,000 inhabitants led to improvements in locomotor function, measured through sarcopenia parameters, and enhanced quality of life in areas such as vitality, mental health, and social functioning. A distinctive feature of this approach is shared decision-making between residents and policymakers, ensuring that solutions are adapted to local realities. This fosters greater adherence, empowerment, and long-term sustainability of co-created strategies.

This project is directly relevant to public policy through collaboration with the Consell Comarcal del Priorat, which represents 23 municipalities. Their recent report identified ageing as a major concern for both institutions and residents. The project's results can therefore guide health policies-decisions, plans, and actions-that address local needs while considering available resources and ensuring long-term sustainability.

By focusing on health promotion and disease prevention, the project ensures that policies are evidence-based and subject to evaluation. The partnership with the Consell Comarcal also aligns with Sustainable Development Goal 3 (Health and Well-being) of the 2030 WHO Agenda and supports the "Health in All Policies" approach, fostering integrated strategies across sectors.

The principal aim of the study is to evaluate the effectiveness of a participatory science intervention study in improving lifestyle habits (dietary habits, physical activity, substance use, and sleep quality), quality of life, emotional well-being, and locomotor capacities through the assessment of sarcopenia parameters (muscle strength, muscle mass, and physical function) in young-old adults (≥60 years) living in rural areas of the Priorat region (Catalonia, Spain).

Specific Objectives:

1. To describe the health status of older people residing in the Priorat region by evaluating: lifestyle habits (diet, substance use, physical activity, and sleep), risk of malnutrition, functional capacity based on sarcopenia parameters, mental capacity (mental health and emotional well-being), and quality of life.
2. To improve lifestyle habits (diet, physical activity, sedentary behaviour, sleep habits, and substance use-alcohol and smoking), emotional well-being and personal relationships to avoid unwanted loneliness, quality of life, and locomotor abilities based on sarcopenia parameters (muscle strength, muscle mass, and physical function).
3. To reduce the risk of malnutrition.
4. To compare the health status of two groups: those aged 60-74 (young-old adults) and those aged 75 and over (older people).
5. To identify the needs, barriers, and motivations of older people through focus groups, including participants aged 60-74, those over 75, and stakeholders such as members of the public administration supporting the project.
6. To compare the differences in needs, barriers, and motivations identified by the young-old adults (60-74 years) and the older people (≥75 years).
7. To actively involve older participants in the co-creation of health promotion activities and an intervention designed for them and their peers.
8. To implement an intervention based on proposals generated during the co-creation process to improve their lifestyle (dietary habits, physical activity, substance use, well-being, and sleep behaviours), quality of life, and locomotor abilities.
9. To analyse environmental barriers, using the "Age-Friendly Cities and Communities Questionnaire (AFCCQ)", in the villages of the Priorat region that may influence the ability to maintain a healthy lifestyle and quality of life for people aged 60-74 and those aged 75 and over.

DETAILED DESCRIPTION:
The study will last for 24 months and will be structured into various tasks:

Tasks 1 and 2. Recruitment of villages and participants

1. Villages: In collaboration with the Consell Comarcal del Priorat, the strategy for contacting the villages will be decided, whether through local councils, community centres, elderly associations, etc. Dissemination may be carried out through posters, social media, letters to residents, electronic bulletins (e-bando), etc.

   The villages in the Priorat region interested in participating will be randomly assigned into two groups: control group (at least 5 villages with 8 participants each) and intervention group (at least 5 villages with 8 participants each).
2. Participants:

   * Older adults (both young-old and elderly) who choose to take part in the project will sign an informed consent form.
   * Stakeholders from the quadruple helix model: companies, government officials, academic institutions, and the community members who may influence the lifestyles of older adults (both young-old adults and elderly) in the rural Priorat region will be contacted by phone or email and informed about the project. Stakeholders will also sign an informed consent form.

Task 3. Characterisation of participants Questionnaires about lifestyles and anthropometric measurements will be completed in small sessions, individually, in person, and on paper. Also, focus groups will be done to gather insights into participants' perceptions of ageing, their needs, barriers, and motivations to improve and maintain healthy lifestyles. Three separate focus groups will be conducted with: young-old adults (60-74 years), elderly adults (≥75 years), and stakeholders, each consisting of 6-8 participants.

Focus groups are structured, moderated group discussions where participants are encouraged to freely express their opinions in response to specific questions. Each session will last approximately 75 minutes and be led by an external moderator.

Baseline data (questionnaires and focus group data) will be analyzed to prepare the co-creation process, ensuring that it is adapted to the real needs and characteristics of the population.

Task 4. Co-creation of solutions Based on the information gathered during the initial characterisation (baseline assessments and focus groups), solutions will be developed through a co-creation process involving older participants (young-old and elderly) from the intervention groups and the stakeholders.

The co-creation session (lasting 4 hours) will follow the PRODUCES framework: a) Problem: Unhealthy lifestyles among people aged ≥ 60 years old, b) Objective: To design solutions to improve lifestyles of people aged ≥ 60 years old, c) Design: Participatory research to increase individual empowerment, d) Users: People aged ≥ 60 years old, e) Co-creators: Stakeholders and older adults, f) Evaluation: Through comparison of intervention and control group, g) Scalability: Model generalisable to other similar areas with elderly populations.

The co-creation process is structured as follows: a) Co-ideation: Word Café dynamics, b) Co-design of the most voted ideas, c) Collaborative prototyping and testing. After sharing ideas, activities, events, dissemination materials, and any other elements deemed necessary to address identified barriers and needs related to lifestyle will be designed.

Proposed activities that provide solutions and fall within the project's budget (agreed upon with the Consell Comarcal del Priorat to ensure sustainability) will be presented and discussed among participants. Finally, participants will take part in prioritizing proposals and defining the final solutions to be implemented."

Task 5. Implementation of the intervention in the intervention villages The co-created intervention for older adults (young-old and elderly) in Priorat villages will be implemented in IG village over 6 months.

Once the intervention has been implemented in intervention villages, the same will be offered to control villages, but without further evaluation, to avoid bias and ensure fair access to potential benefits.

Task 6. Participant characterization (younger-old and older-old) - final assessment: Both participants who received the intervention and those in the control group will be evaluated by questionnaires about lifestyles and anthropometric measurements, to compare any differences between those who underwent the intervention and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Signed informed consent
* Living independently
* Capacity to follow and complete the study
* Resident in one of the villages of the Priorat region

Exclusion Criteria:

Failure to meet any of the inclusion criteria will be considered grounds for exclusion.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional intake | Baseline and follow-up (6 months later)
  The Food Frequency Consumption Questionnaire (FFCQ) (Rodríguez IT, et al. Nutr Hosp. 2008) to assess the nutritional intake of elderly participants.
Physical activity and sedentary behaviour | Baseline and follow-up (6 months later)
  International physical activity questionnaire for elderly: IPAQ for elderly IPAQ-E, Spanish version (Rubio-Castañeda et al., 2017). Higher scores mean a better outcome.
Sleep quality | Baseline and follow-up (6 months later)
  Pittsburgh questionnaire (Buysse et al., 1989). The maximum score is 21 points. More than 5 points are considered bad outcomes and sleep problems, and less than 5 points are considered better outcomes and no sleep problems.
Depressive symptoms | Baseline and follow-up (6 months later)
  Geriatric Depression Scale Questionnaire (Yesavage et al., 1983). The maximum punctuation is 15. The score is 0-4, no depression; 5-8, mild depression; 9-11, moderate depression; and 12-15, severe depression.
Quality of life behaviours | Baseline and follow-up (6 months later)
  Quality of life assessed by the SF-36 Health survey questionnaire (Ware & Sherbourne, 1992) and the EuroQol-5D questionnaire (Herdman M et al., 2001). Higher scores mean a better outcome.
Muscle strength | Baseline and follow-up (6 months later)
  The muscle strength assessed by handgrip dynamometry (Jamar dynamometer; Sammons Preston Rolyan, Bolingbrook, IL).
Muscle mass | Baseline and follow-up (6 months later)
  Muscle mass (appendicular skeletal muscle mass (kg)) assessed by Bioimpedance TANITA (MC-780MA; Tanita Corp., Tokyo, Japan).
Physical performance | Baseline and follow-up (6 months later)
  Gait speed (m/s) assessed by the length of the walking course divided by the time (Ladang et al., 2023).
Nutritional status | Baseline and follow-up (6 months later)
  Hemoglobin (g/dl) in blood samples assessed by HemoCue® Hb 801 (HemoCue AB, Ängelholm, Suecia, 2020).

SECONDARY OUTCOMES:
Nutritional status | Baseline and follow-up (6 months later)
  Mini Nutritional Assessment Short-Form (MNA-SF). The maximum punctuation is 14 points. The score is 0-7 points (malnutrition), 8-11 points (risk of malnutrition), and 12-14 points (normal nutritional status).
Anthropometric measures | Baseline and follow-up (6 months later)
  Height (cm) measured by wall-mounted stadiometer (Tanita Leicester Portable; Tanita Corp., Barcelona, Spain)
Anthropometric measures | Baseline and follow-up (6 months later)
  Weight (kg) measured by calibrated scale (TANITA MC-780MA; Tanita Corp., Tokyo, Japan).
Anthropometric measures | Baseline and follow-up (6 months later)
  BMI (kg/m2) is calculated by dividing weight (kg) by height (m2).
Anthropometric measures | Baseline and follow-up (6 months later)
  WC: waist circumference (cm) measured by steel measuring tape (at the umbilicus).
Anthropometric measures | Baseline and follow-up (6 months later)
  Calf circumference(cm) measured by steel measuring tape.
Vascular parameters | Baseline and follow-up (6 months later)
  Systolic and diastolic blood pressure (SBP and DBP) (mm Hg) and pulse pressure (PP) (mm Hg) assessed by an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Muscle mass | Baseline and follow-up (6 months later)
  Muscle mass thickness of quadriceps and forearm assessed by ultrasound (VINNO 5 (Vinno (Suzhou) Co., Ltd., China)
Abdominal fat | Baseline and follow-up (6 months later)
  Abdominal fat assessed by ultrasound (VINNO 5 (Vinno (Suzhou) Co., Ltd., China)
Healthy and friendly communities | Baseline and follow-up (6 months later)
  Age-Friendly Cities and Communities Questionnaire (AFCCQ) with eight domains (housing, social participation, respect and social inclusion, civic participation and employment, communication and information, community support and health services, outdoor spaces and buildings, transportation, financial situation). All domains are answered on a 5-point scale, ranging from totally disagree to totally agree. Scores: -2 = totally disagree; -1 = disagree; 0 = neutral; 1 = agree; 2 = totally agree. Higher scores in each domain mean a better outcome.
Socio-familiar situation | Baseline and follow-up (6 months later)
  Socio-familiar situation assessed through the validated questionnaire Socio-Familial Assessment Scale (TSO) (Giménez Bertomeu VM, et al. 2020), based on different indicators (family structure and function, social contacts, required support, and receipt of resources for activities of daily living, economic income, and housing).
Other health determinants | Baseline and follow-up (6 months later)
  Other health determinants that participants considered important to address, selected during the focus groups.
Lipid profile | Baseline and follow-up (6 months later)
  Total cholesterol (mmol/L) in blood samples assessed by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Lipid profile | Baseline and follow-up (6 months later)
  HDLc (mmol/L) in blood samples assessed by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Lipid profile | Baseline and follow-up (6 months later)
  LDLc (mmol/L) in blood samples assessed by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Lipid profile | Baseline and follow-up (6 months later)
  Total TG (mmol/L) in blood samples assessed by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Glucose homeostasis | Baseline and follow-up (6 months later)
  Fasting blood glucose (mmol/L)in blood samples assessed by OneTouch Select Plus Flex®.
Glucose homeostasis | Baseline and follow-up (6 months later)
  HGBA1c (%) in blood samples assessed by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Inflamation markers | Baseline and follow-up (6 months later)
  High-sensitivity C-reactive protein (mg/dL) in blood samples assessed by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Urine metabolites | Baseline and follow-up (6 months later)
  Metabolomic characterization: targeted metabolomics for the detection of over 1,000 metabolites. Targeted metabolomic analysis is performed using a liquid chromatography-tandem mass spectrometry (LC-MS/MS) platform, employing multiple reaction monitoring (MRM) in both positive and negative ionization modes. The protocol includes a prior chemical derivatization step, followed by separation via reversed-phase liquid chromatography (RP-LC) and/or direct flow injection to the mass spectrometer (DFI-MS) for the analysis of the target metabolites. Quantification is carried out using internal isotopic standards and multipoint calibration curves, allowing for absolute concentration determination. (Zheng J, et al. Anal Chem. 2020; 92(15):10664-70/ Zhang L, et al. Metabolites. 2024;14(11):622)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Rovira i Virgili, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No